CLINICAL TRIAL: NCT01405417
Title: Endoscopic Peroral Myotomy for Treatment of Achalasia: Multicenter Study
Brief Title: Endoscopic Peroral Myotomy for Treatment of Achalasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough data collected
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Prof. Dr. Thomas Roesch, Universitätsklinikum Hamburg-Eppendorf, Endoscopy department, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKE HH Endoscopy PV3725mc
Record Dates: First submitted 2011-05-26; First posted 2011-07-29 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Achalasia
Keywords: Achalasia; Heller myotomy; Dysphagia; Peroral Endoscopic Myotomy
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peroral endoscopic myotomy (Experimental): Patients with achalasia who are designed to either have balloon dilatation or botulinum toxine injection, or to have surgical intervention (Heller myotomy) for therapy.
  Peroral endoscopic myotomy: A forward-viewing upper endoscope is used with a transparent distal cap attachment. Carbon dioxide gas is necessary for insufflation during the procedures. An endoscopic knife is used to access the submucosa, dissect the submucosal tunnel and also to divide circular muscle bundles over a length of approximately 10cm, extending 2-3cm onto the cardia. A electrogenerator is used with spray coagulation mode. A coagulating forceps is used for hemostasis as needed. Closure of the mucosal entry site is performed using standard endoscopic clips.
  Interventions: Procedure: Endoscopic Peroral Myotomy

INTERVENTIONS:
Procedure: Endoscopic Peroral Myotomy — Endoscopic peroral myotomy: A forward-viewing upper endoscope is used with a transparent distal cap attachment. Carbon dioxide gas is necessary for insufflation during the procedures. An endoscopic knife is used to access the submucosa, dissect the submucosal tunnel and also to divide circular muscle bundles over a length of approximately 10cm, extending 2-3cm onto the cardia. A electrogenerator is used with spray coagulation mode. A coagulating forceps is used for hemostasis as needed. Closure of the mucosal entry site is performed using standard endoscopic clips.

SUMMARY:
This study intends to investigate the feasibility, safety and efficacy of peroral endoscopic myotomy for the treatment of achalasia in a multi center setting.

DETAILED DESCRIPTION:
This study intends to investigate the feasibility, safety and efficacy of peroral endoscopic myotomy for the treatment of achalasia in a multi center s

70 patients will be enrolled to evaluate feasibility, safety and efficacy of peroral endoscopic myotomy. Main outcome measurement is the Eckardt symptom score at 3 month after peroral endoscopic myotomy.

Primary outcome:

-Eckhard symptom score 3 month after therapy.

Secondary outcomes:

Lower esophageal sphincter pressure at 3 month after therapy. Reflux symptoms at 3 month after therapy. For this prospective study, inclusion criteria are achalasia, as diagnosed by established methods (contrast fluoroscopy, manometry, esophago-gastro-duodenoscopy) and age greater than 18 years. Previous therapy, such as esophageal surgery or previous myotomy are exclusion criterion.

A forward-viewing upper endoscope is used with a transparent distal cap attachment. Carbon dioxide gas is necessary for insufflation during the procedures. An endoscopic knife is used to access the submucosa, dissect the submucosal tunnel and also to divide circular muscle bundles over a length of approximately 10cm, extending 2-3cm onto the cardia. A electrogenerator is used with spray coagulation mode. A coagulating forceps is used for hemostasis as needed. Closure of the mucosal entry site is performed using standard endoscopic clips.

ELIGIBILITY:
Inclusion Criteria:

* Patient with symptomatic achalasia and pre-op barium swallow, manometry and esophagogastroduodenoscopy which are consistent with the diagnosis
* persons of age > 18 years with medical indication for surgical myotomy or Endoscopic balloon dilatation
* Signed written informed consent.

Exclusion Criteria:

* Patients with previous surgery of the stomach or esophagus
* Patients with known coagulopathy
* Previous achalasia-treatment with surgery
* Patients with liver cirrhosis and/or esophageal varices
* Active esophagitis
* Eosinophilic esophagitis
* Barrett's esophagus
* Pregnancy
* Stricture of the esophagus
* Malignant or premalignant esophageal lesion
* Candida esophagitis
* Hiatal hernia > 2cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Eckhard symptom score at 3 month after peroral endoscopic myotomy | Score is evaluated at 3 month after peroral endoscopic myotomy
  Validated symptom score based on dysphagia, pain, regurgitation and weight loss

SECONDARY OUTCOMES:
Lower esophageal sphincter pressure | Lower esophageal sphincter pressure is determined by manometry at 3 month after peroral endoscopic myotomy
  Manometry study
Reflux Symptoms | Reflux Symptoms are evaluated at 3 month after peroral endoscopic myotomy
  Symptoms as reported by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roesch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Clinic for Visceral- and Thoracic Surgery, McGill University Health Centre, Montreal, Quebec, Canada
- Germany (2):
  - Clinic for Visceral-, Vasular- and Thoracic Surgery, Markus-Krankenhaus, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Interdisziplinäre Endoskopie, Hamburg
- Department of Gastroenterology and Hepatology, Academic Medical Center, Amsterdam, Netherlands
- Klinik für Gastroenterologie, USZ, Zurich, Switzerland

REFERENCES:
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Result] Von Renteln D, Fuchs KH, Fockens P, Bauerfeind P, Vassiliou MC, Werner YB, Fried G, Breithaupt W, Heinrich H, Bredenoord AJ, Kersten JF, Verlaan T, Trevisonno M, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: an international prospective multicenter study. Gastroenterology. 2013 Aug;145(2):309-11.e1-3. doi: 10.1053/j.gastro.2013.04.057. Epub 2013 May 9. PMID 23665071
- [Result] Werner YB, Costamagna G, Swanstrom LL, von Renteln D, Familiari P, Sharata AM, Noder T, Schachschal G, Kersten JF, Rosch T. Clinical response to peroral endoscopic myotomy in patients with idiopathic achalasia at a minimum follow-up of 2 years. Gut. 2016 Jun;65(6):899-906. doi: 10.1136/gutjnl-2014-308649. Epub 2015 Apr 30. PMID 25934759
- [Result] Werner YB, von Renteln D, Noder T, Schachschal G, Denzer UW, Groth S, Nast JF, Kersten JF, Petzoldt M, Adam G, Mann O, Repici A, Hassan C, Rosch T. Early adverse events of per-oral endoscopic myotomy. Gastrointest Endosc. 2017 Apr;85(4):708-718.e2. doi: 10.1016/j.gie.2016.08.033. Epub 2016 Sep 5. PMID 27609778
- [Derived] Nast JF, Berliner C, Rosch T, von Renteln D, Noder T, Schachschal G, Groth S, Ittrich H, Kersten JF, Adam G, Werner YB. Endoscopy versus radiology in post-procedural monitoring after peroral endoscopic myotomy (POEM). Surg Endosc. 2018 Sep;32(9):3956-3963. doi: 10.1007/s00464-018-6137-9. Epub 2018 Mar 15. PMID 29546671
- [Derived] Verlaan T, Ponds FA, Bastiaansen BA, Bredenoord AJ, Fockens P. Single clips versus multi-firing clip device for closure of mucosal incisions after peroral endoscopic myotomy (POEM). Endosc Int Open. 2016 Oct;4(10):E1052-E1056. doi: 10.1055/s-0042-113126. Epub 2016 Sep 21. PMID 27747277
- See also: University Hospital Hamburg-Eppendorf, Endoscopy Department — http://www.uke.de/kliniken/endoskopie/index.php